CLINICAL TRIAL: NCT06189378
Title: Picture This: A Randomized Controlled Pilot Study Investigating Adherence to Blood Pressure Diaries With Personalized Visuals
Brief Title: Adherence to Blood Pressure Diaries With Personalized Visuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Clemens Farr, MD PhD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1249/2023
Record Dates: First submitted 2023-12-08; First posted 2024-01-03 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Neurovascular Disorder
Keywords: adherence; blood pressure diary; stroke; TIA
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional blood pressure diary (Active Comparator): Blood pressure diaries consisted of tables including columns for date, time as well as systolic and diastolic blood pressure respectively (1 page for 1 week) printed on the right-hand pages of an A5 (ISO 216 format) booklet.
  Interventions: Other: Conventional blood pressure diary
- Blood pressure diary including patient-provided pictures (Experimental): In the interventional arm pictures chosen by patients were provided over a secure online connection by patients in this group and inserted into the left-hand-pages of the blood pressure diaries.
  Interventions: Other: Inclusion of patient-provided pictures into blood pressure diaries

INTERVENTIONS:
Other: Inclusion of patient-provided pictures into blood pressure diaries — Patient-provided pictures with positive meaning were included into blood pressure diaries
  Arms: Blood pressure diary including patient-provided pictures
Other: Conventional blood pressure diary — Conventional blood pressure diary
  Arms: Conventional blood pressure diary

SUMMARY:
This trial randomizes patients with a neurovascular diagnosis to a type of blood pressure diary for secondary stroke prevention (conventional blood pressure diary or blood pressure diary including patient-provided images). Outcomes include adherence and patient-reported outcomes.

DETAILED DESCRIPTION:
In this prospective trial, the investigators randomized persons with diagnoses of stroke or transitoric ischemic attack into two groups: (i) 10 patients received a personalized blood pressure diary with pictures of their choosing. (ii) 10 patients received a blood pressure diary without photographs. The investigators instructed participants in either group to document their blood pressure at home twice daily over twenty-eight days.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of TIA or stroke (ischemic or hemorrhagic) upon admission.

Exclusion Criteria:

* Modified Rankin Scale score of ≥4 at inclusion
* Inability to provide informed consent
* Pre-existing legal guardianship.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Adherence | 28 days
  The primary endpoint was adherence to blood pressure diaries defined as the number of complete blood pressure measurements (maximum of two per day) divided by the maximum number of measures over the study period (28 days, resulting in a maximum total of 56 measurements). Complete entries were defined as diary entries stating date, time and systolic as well as diastolic blood pressure.

SECONDARY OUTCOMES:
Blood pressure | 28 days
  Mean raw values of systolic and diastolic blood pressure
Precision of documentation of blood pressure | 28 days
  The proportion of documented values ending with "0" or "5" served to assess the extent of rounding (i.e. the precision of documentation)
Patient Global Impression of Change Scale | 28 days
  The Patient Global Impression of Change Scale is a self-report rating scale of 1 item on a Likert scale (maximum 7, higher score is better) and 1 item on a scale from 0-10 (higher score is worse). It was applied to assess patient satisfaction.
36-Item Short Form Health Survey | 28 days
  The 36-Item Short Form Health Survey is a self-report survey of items on a Likert Scale in 8 domains. It is designed to assess quality of life. The maximum amount of points is 100. More points are better.
Hospital Anxiety and Depression Scale | 28 days
  The Hospital Anxiety and Depression Scale is a self-report rating scale of 14 items on a Likert scale. It is designed to measure anxiety and depression (7 items for each subscale). The maximum amount of points in each subscale is 21. More points are worse.

OTHER OUTCOMES:
Exploratory endpoints | 28 days
  Exploratory endpoints evolved around patients' perspectives on blood pressure diaries as assessed by an empirical survey (13 questions in each group) conceived for this study. Possible answers were Likert-type scales, yes/no or open commentaries.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Farr, MD PHD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request and through our local ERB.
Supporting Information: Study Protocol, ICF
Time Frame: Upon request and for 1 month
Access Criteria: reasonable request and upon approval of our local ERB